CLINICAL TRIAL: NCT06645522
Title: Safety and Efficacy of Edaravone Dexborneol for Acute Ischemic Stroke: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Safety and Efficacy of Edaravone Dexborneol for Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Vice President of the First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ED-AIS
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Edaravone Dexborneol
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edaravone dexborneol group (Experimental): Edaravone dexborneol injection 37.5mg every 12 hours for 7 days and a sublingual dose of edaravone dexborneol 36 mg twice a day for 21 days.
  Interventions: Drug: Edaravone dexborneol
- Placebo group (Placebo Comparator): Placebo injection every 12 hours for 7 days and a sublingual dose of placebo drug twice a day for 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Edaravone dexborneol — Edaravone dexborneol injection 37.5mg (edaravone 30mg and dexborneol 7.5mg) and 100ml of 0.9% saline every 12 hours for 7 days; sequentially a sublingual dose of edaravone dexborneol 36 mg (edaravone, 30 mg; dexborneol, 6 mg) twice a day for 21 days.
  Arms: Edaravone dexborneol group
Drug: Placebo — Placebo injection every 12 hours for 7 days; sequentially a sublingual dose of placebo drug twice a day for 21 days.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine the efficacy and safety of edaravone dexborneol in treating acute ischemic stroke.

DETAILED DESCRIPTION:
In this study, 1200 patients with acute ischemic stroke within 48 hours from the onset are included in several centres in China according to the principles of randomization, double-blind, and parallel control. The experimental group receives basic treatment and edaravone dexborneol injection for 7 consecutive days, and sequentially receives a sublingual dose of edaravone dexborneol for 21 consecutive days. The placebo group receives basic treatment and edaravone dexborneol placebo injection for 7 consecutive days and sequentially receives a sublingual dose of edaravone dexborneol placebo drug for 21 consecutive days. Two groups will be followed up at day 90 to evaluate the efficacy and safety of edaravone dexborneol in treating acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 80 years old, regardless of gender;
2. Patients diagnosed as acute ischemic stroke according to "key points for diagnosis of all kinds of major cerebrovascular diseases in China 2019", and able to randomise and initiate edaravone dexborneol treatment less than or equal to 48 hours of stroke onset.
3. Total National Institute of Health stroke scale (NIHSS)≥6 and ≤24, and the sum of NIHSS score for the upper limb and the lower limb is greater than or equal to 2;
4. modified Rankin Scale (mRS) score of 1 or less before onset.
5. Did not receive edaravone dexborneol treatment before enrollment;
6. The informed consent approved by the ethics committee was voluntarily signed by the patient or his legal representative.

Exclusion Criteria:

1. Reperfusion therapy (intravenous thrombolysis and endovascular therapy) has been received or planned after stroke onset.
2. Transient ischemic attack (TIA);
3. Posterior circulation stroke;
4. Intracranial hemorrhagic diseases seen in head imaging: hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc;
5. Severe disturbance of consciousness: the item score of 1a consciousness level of NIHSS was more than 1;
6. Patients with severe mental disorders and dementia;
7. Systolic blood pressure after blood pressure control is still higher than 220mmhg or diastolic blood pressure was higher than 120mmhg;
8. Severe cardiac insufficiency, dissection and acute pericarditis; Severe liver insufficiency, ALT or AST > 3.0 × ULN; Or severe active liver diseases have been diagnosed, such as acute hepatitis, chronic active hepatitis, cirrhosis, etc;Severe renal insufficiency, Serum Creatinine (SCr) is greater than 200μmol/L, Creatinine Clearance (CrCl) is less than 30 ml/min or receiving hemodialysis; Or suffering from severe systemic diseases, the estimated survival time is less than 90 days;
9. Complicated with malignant tumor or undergoing anti-tumor treatment;
10. Therapeutic neuroprotective agents have been applied after onset of stroke, including commercially available edaravone, nimodipine, ganglioside, citicoline, piracetam, butyl benzene peptides, Urinary Kallidinogenase, Ginkgolide.
11. Patients during pregnancy, lactation and planned pregnancy;
12. Allergic to dexborneol or edaravone or excipients;
13. Have participated in other clinical studies or are participating in other clinical studies within 30 days before randomization;
14. Patients who are unwilling to be followed up，and the investigators consider the patients are not suitable for this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
modified rankin scale (mRS) score ≤ 1 | Day 90 after randomization
  The proportion of patients with mRS score of 1 or less on day 90 after randomization. Ranged from 0 to 6, a low value represents a better outcome.

SECONDARY OUTCOMES:
Serum ubiquitin C-terminal hydrolase L1 (UCH-L1), glial fibrillary acidic protein (GFAP), S100β, neuron-specific enolase (NSE) levels | Day 3 after randomization
Serum ubiquitin C-terminal hydrolase L1 (UCH-L1), glial fibrillary acidic protein (GFAP), S100β, neuron-specific enolase (NSE) levels | Day 7 after randomization
NIHSS score on day 7 | Day 7 after randomization
  NIHSS (National Institute of Health stroke scale) score on day 7 after randomization. NIHSS ranged from 0 to 42, a low value represents a better outcome.
mRS score ≤ 2 | Day 90 after randomization
  The proportion of patients with an mRS score of 2 or less on day 90 after randomization. Ranged from 0 to 6, a low value represents a better outcome.
Distribution of mRS score | Day 90 after randomization
  Distribution of modified Rankin score on day 90 after randomization. Ranged from 0 to 6, a low value represents a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China